CLINICAL TRIAL: NCT03182452
Title: Outcomes and User Acceptance of the IntelliVue Alarm Advisor Software (Europe)
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: PMS-BBN-EU-AA-1.00
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Clinical Alarms
Keywords: Alarms; Alarm Fatigue; Alarm Nuisance; Alarm Reduction; Patient Monitoring; Intensive Care
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Pre Phase (no Alarm Advisor): No Software installed
- Post Phase (Alarm Advisor installed): Software implemented and staff trained (Interventional Phase)
  Interventions: Other: Alarm Advisor

INTERVENTIONS:
Other: Alarm Advisor — Providing advice on alarm limits as part of routine medical care
  Groups: Post Phase (Alarm Advisor installed)

SUMMARY:
This Clinical Study will be conducted as a comparative study focusing on usability and efficiency by comparing alarm burden pre- and post-implementation of an "Alarm Advisor software".

DETAILED DESCRIPTION:
In a first phase of data collection (pre-implementation) all alarms of an intensive care unit population are recorded.

In an interim period an Alarm Advisor software will be introduced to the unit.

In a second phase (post-implementation) the same set of alarm data will be recorded.

The "Alarm Advisor" Software can identify alarms based on criteria set by the medical staff and provide hints to reduce alarms and alarm nuisance (e.g. by proposing adjustments of alarm limits).

The effect of reduction of recurring nuisance alarms through the implementation of the Alarm Advisor shall be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit during the study period

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Monitored intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 1487 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Clinical Alarms | six to eight months
  Number of Different Alarms on Intensive Care

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trick, MD, Principal Investigator — Klinikum Konstanz, Germany
Locations (1):
- Klinikum Konstanz, Konstanz, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No